CLINICAL TRIAL: NCT06700213
Title: Guideline Directed Medical Therapy in Patients With Heart Failure
Acronym: TEAM-MGH
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, James L. Januzzi, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2023P001526
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: heart failure; quality improvement; angiotensin converting enzyme inhibitors; angiotensin receptor/neprilysin inhibitors; angiotensin II receptor blockers; evidence based beta blockers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample for circulating biomarkers is obtained at baseline and as part of routine follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Heart Failure: Cohort will be comprised of a minimum of 75 participatns with HFrEF and a minimum of 25 participants with HFmrEF/HFpEF. At each visit, presence of intolerances to GDMT will be sought and recorded. Medications will include those outlined by GDMT, including angiotensin receptor/neprilysin inhibitors (ARNI), angiotensin II receptor blockers (ARB), angiotensin converting enzyme inhibitors (ACEi), evidence based beta blockers (eBBB), aldosterone receptor antagonists (MRA), and sodium-glucose co-transporter 2 (SGLT2) inhibitors.
- Research Patient Data Repository (RPDR): Patients will be selected from those with available data following May of 2020 (after regulatory approval of SGLT2 inhibitors for treatment of HFrEF) or in the case of HFpEF following February 2022.

SUMMARY:
The TEAM-MGH study will formerly evaluate impact of the GDMT Clinic versus matched usual care patients on the proportion of GDMT administration over a 12 week period in approximately 300 total patients with HF across the spectrum of LVEF (with a minimum of 150 with HFrEF). The study will also assess impact of the GDMT Clinic on health status, functional capacity, biomarker profiles, cardiac remodeling and cardiovascular events.

DETAILED DESCRIPTION:
The lack of adherence to Goal-Directed Medical Therapy (GDMT) is a major problem in modern HF care. Despite advances in therapies for those with HF along with well-articulated goals for achieving guideline-directed medical therapy (GDMT) for affected individuals, the treatment of persons with HF lags behind current recommended guideline approaches, with 30% of ambulatory patients with HFrEF not being prescribed angiotensin receptor/neprilysin inhibitors (ARNI), angiotensin converting enzyme inhibitors (ACEi), angiotensin II receptor blockers (ARB), or evidence based beta blockers (eBBB) and the majority not receiving target doses of these medications despite lack of medical contraindications. The reasons for gaps in care include hesitancy to change medical programs in ostensibly stable patients, concerns about risk of drug intolerances, worries about drug costs, as well as uncertainty about benefits. Additionally, complexity of medical therapy, rapid evolution in the currently recommended therapeutic options, and challenges in care coordination also result in missed treatment opportunities. Given that most individuals with HF are cared for by specialists other than those trained in advanced HF therapies, this intersection of increasing complexity of care results in substantial gaps in care. The proposed research is to study impact of the GDMT clinic for patients across the spectrum of HF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HF, including new onset disease
* Established cardiovascular follow up at MGH
* Receiving sub-optimal medical care defined as <50% target doses of GDMT agents
* Age ≥18 years
* For HFpEF:

  * Presence of structural heart disease (LAVi >34 mL/Kg2, E/e' >14, or LVH)
  * Recent HF hospitalization or historical NT-proBNP >300 pg/mL

Exclusion Criteria:

* Planned referral to the Advanced HF program
* Decompensated HF
* End-stage kidney disease

  * eGFR <15 mL/min/1.73m2 or on renal replacement therapy
* Untreated severe valvular heart disease
* Advanced HF

  * Inotropic support
  * Transplant or MCS planned
  * Enrolled in hospice or palliative care
* Life expectancy <12 months due to non-CV disease
* Pericardial constriction
* Hypertrophic cardiomyopathy
* Unwillingness or inability to take GDMT
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients with NYHA Class I-IV HF, aged ≥18 years, directly referred to GDMT Clinic from cardiology clinics at MGH. A minimum of 75 patients with HFrEF will be included in the GDMT Clinic arm. Patients with improved EF will be included as HFrEF.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
GDMT Administration for HF | 12 weeks
  Effect of GDMT Clinic versus Usual Care on administration of GDMT for HF.

SECONDARY OUTCOMES:
Mechanistic HF Outcomes | 12 weeks
  Effect of GDMT Clinic versus Usual Care on changes in mechanistic HF outcomes.

OTHER OUTCOMES:
Tolerability of GDMT Initiation | 12 weeks
  Assess tolerability of rapid-sequence initiation of GDMT in the GDMT Clinic
Outcomes at 6 Months | 6 months
  Effect of GDMT Clinic versus Usual Care on incident cardiovascular outcomes during a 6 month follow up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spahillari A, Cohen LP, Lin C, Liu Y, Tringale A, Sheppard KE, Ko C, Khairnar R, Williamson KM, Wasfy JH, Scott NS, Paquette C, Greene SJ, Fonarow GC, Januzzi JL Jr. Efficacy, Safety and Mechanistic Impact of a Heart Failure Guideline-Directed Medical Therapy Clinic. JACC Heart Fail. 2025 Apr;13(4):554-568. doi: 10.1016/j.jchf.2024.08.017. Epub 2024 Oct 9. PMID 39387769